CLINICAL TRIAL: NCT04291326
Title: A Study on Cerebral Blood Flow Velocity Changes During Laparoscopic Surgery in Pediatric Patients: Observational Study Using Transfontanelle Ultrasound
Brief Title: Cerebral Blood Flow Velocity Changes During Laparoscopic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Other Study IDs: 2002-036-110
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Blood Flow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transfontanelle ultrasound — cerebral blood flow measurement using transfontanelle ultrasound

SUMMARY:
Little is known about how implementation of pneumoperitoneum contributes to cerebral blood flow in pediatrics. We investigated this question in patients undergoing laparoscopic surgery, hypothesizing that cardiorespiratory changes during this procedure would reduce cerebral perfusion.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing laparoscopic surgery

Exclusion Criteria:

-

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients undergoing general anesthesia for laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | intraoperative
  cerebral blood flow measurement using transfontanelle ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided